CLINICAL TRIAL: NCT05220826
Title: Early eNdovascular Embolization for Chronic subduraL hematOma After SUrgery and Prevention of REcurrence (ENCLOSURE)
Brief Title: Endovascular Embolization of Chronic Subdural Hematomas After Surgery
Acronym: ENCLOSURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)575/2021
Record Dates: First submitted 2022-01-04; First posted 2022-02-02 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Chronic Subdural Hematoma
Keywords: Middle meningeal artery embolization
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Ethanol; ethylene-vinyl alcohol copolymer; Dimethyl Sulfoxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Primary outcome will be assesed by a blinded external core lab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical drainaje (the standar of care) (No Intervention): Surgery will consist of performing a craniotomy (burr hole or drill) and evacuation of the hematoma. Depending on the operator, the surgical procedure may incorporate the use of subdural space drainage devices (e.g. Jackson Pratt drainage) connected to a soft suction reservoir. If used, these devices should be removed within 48 hours of installation.
- Surgical drainaje plus early embolization of middle meningeal artery (Experimental): The endovascular procedure will be performed until 72 hours after surgical evacuation of chronic subdural hematoma. Embolization will be performed with non-adhesive embolizing fluids such as Onix®, Phil®, Squid® or Libro®.
  Interventions: Procedure: Post surgical embolization of middle meningeal artery with liquid embolic agents (ethylene vinyl alcohol copolymers as Onix, Squid, Phil or Libro)

INTERVENTIONS:
Procedure: Post surgical embolization of middle meningeal artery with liquid embolic agents (ethylene vinyl alcohol copolymers as Onix, Squid, Phil or Libro) — The endovascular procedure will be performed until 72 hours after surgical evacuation of chronic subdural hematoma. Embolization will be performed with non-adhesive embolizing fluids such as Onix®, Phil®, Squid® or Libro®.
  Other Names: Liquid embolic agent: Onix (ethylene vinyl alcohol copolymer), Medtronic.; Liquid embolic agent: Squid (ethylene vinyl alcohol copolymer), Balt.; Liquid embolic agent: Phil (copolymer disolved in DMSO), Microvention-Terumo.; Liquid embolic agent: Libro (ethylene vinyl aalcohol copolymer), Invamed.
  Arms: Surgical drainaje plus early embolization of middle meningeal artery

SUMMARY:
Chronic subdural hematomas (CSH) are one of the most frequent pathologies in emergency neurosurgical practice. Standard therapy for symptomatic CSH is surgical drainage. However, the recurrence rate after surgery is high (10 to 20% in the most of series, although it has been reported from 2 to 37%). Middle meningeal artery embolization (MMAE) is a promising minimally invasive procedure that has recently been proposed as an alternative or adjunctive treatment to surgery. The investigators hypothesize that early post operative endovascular treatment can reduce the recurrence rate in high-risk patients, improving neurological outcomes by reducing the need for reinterventions, hospitalizations, and post-operative complications. The aim of the investigators is to analyze the efficacy of and safety of early post-surgical embolization of MMA in reducing the risk of CSH recurrence.

DETAILED DESCRIPTION:
The study was designed as an open-label, multicenter randomized trial involving patients with symptomatic CSH and surgical evacuation criteria. Patients will be randomized in a 1: 1 ratio to receive surgical drainage (the standard of care) or surgical drainage plus early endovascular embolization of MMA (< 72 hours after surgery). Endovascular procedures will be performed with non-adhesive embolizing fluids. The primary outcome will be the recurrence of CSH at 6 months and secondary outcomes will be the risk reduction of recurrence in patients with risk factors, functional status measured by the modified Rankin scale (range, 0 [no disability] to 6 [death]) at 6 months and complications related to endovascular procedure.

ELIGIBILITY:
Inclusion Criteria:

* Chronic subdural hematoma equal or greater than 10 mm, midline shift equal or greater than 5 mm or neurological symptoms attributable to mass effect.
* Recent diagnosis or recurrence
* Surgical treatment performed < 72 hours
* Informed consent signed by the patient or they responsible family member

Exclusion Criteria:

* Advanced disease with life expectancy < 6 months
* Condition that contraindicated endovascular procedure: Pregnancy, renal failure defined as creatinine clearence < 30 ml/min, allergy to iodinated contrast.
* Unavailability for follow up st 6 months
* Patient expressly refuses treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of chronic subdural hematoma | 6 months
  Defined ad reappearance of symptomatic blood collection or whose thickness is > 1 cm or which determines a deviation from the midline> 5 mm

SECONDARY OUTCOMES:
Functional status | 6 months
  Measured by modified Rankin scale (range, 0 [no disability] to 6 [death])
Safety of endovascular treatment | 6 months
  Measured by complications related to endovascular procedure
Hematoma reabsorption speed | 6 months
  Measured by hematoma volume after treatment on CT imaging
Cumulative days of hospital stay | 6 months
  Measured in both groups (surgical alone and surgical plus endovascular)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Tomasello, MD, Study Chair — Hospital Universitari Vall d'hebron Barcelona, Spain; Jose Luis Cuevas, MD, Principal Investigator — Hospital de Puerto Montt, Puerto Montt, Chile.
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No